CLINICAL TRIAL: NCT02192463
Title: Relative Bioavailability of Different Oral Viramune Extended Release Formulations Containing 300 mg or 400 mg Compared to 200 mg or 400 mg as One or Two 200 mg IR Tablets Following Administration in Healthy Male Volunteers - an Openlabel, Non-randomized, Parallel Group Study
Brief Title: Relative Bioavailability of Different Oral Viramune Extended Release Formulations Compared to Viramune® Oral Suspension in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1100.1485
Record Dates: First submitted 2014-07-15; First posted 2014-07-16 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Healthy
MeSH Terms: interventions — Nevirapine

ARMS (12):
- Nevirapine (NVP) ER 300 mg (KCR 20%) Medium Release (Experimental)
  Interventions: Drug: NVP ER 300 mg (KCR 20%) Medium Release
- NVP ER 300 mg (KCR 25%) Medium Release (Experimental)
  Interventions: Drug: NVP ER 300 mg (KCR 25%) Medium Release
- NVP ER 300 mg (KCR 30%) Slow Release (Experimental)
  Interventions: Drug: NVP ER 300 mg (KCR 30%) Slow Release
- NVP ER 400 mg (KCR 25%) Medium Release (Experimental)
  Interventions: Drug: NVP ER 400 mg (KCR 25%) Medium Release
- NVP ER 300 mg (KCR 40%) Slow Release (Experimental)
  Interventions: Drug: NVP ER 300 mg (KCR 40%) Slow Release
- NVP ER 300 mg (ECR 20%) Fast Release (Experimental)
  Interventions: Drug: NVP ER 300 mg (ECR 20%) Fast Release
- NVP ER 400 mg (KCR 20%) Medium Release (Experimental)
  Interventions: Drug: NVP ER 400 mg (KCR 20%) Medium Release
- NVP ER 400 mg (KCR 30%) Slow Release (Experimental)
  Interventions: Drug: NVP ER 400 mg (KCR 30%) Slow Release
- NVP ER 400 mg (KCR 40%) Slow Release (Experimental)
  Interventions: Drug: NVP ER 400 mg (KCR 40%) Slow Release
- NVP ER 400 mg (ECR 20%) Fast Release (Experimental)
  Interventions: Drug: NVP ER 400 mg (ECR 20%) Fast Release
- Nevirapine IR 1 tablet (Active Comparator)
  Interventions: Drug: Nevirapine immediate release (IR) 200 mg
- Nevirapine IR 2 tablets (Active Comparator)
  Interventions: Drug: Nevirapine immediate release (IR) 200 mg

INTERVENTIONS:
Drug: NVP ER 300 mg (KCR 20%) Medium Release
  Arms: Nevirapine (NVP) ER 300 mg (KCR 20%) Medium Release
Drug: NVP ER 300 mg (KCR 25%) Medium Release
  Arms: NVP ER 300 mg (KCR 25%) Medium Release
Drug: NVP ER 300 mg (KCR 30%) Slow Release
  Arms: NVP ER 300 mg (KCR 30%) Slow Release
Drug: NVP ER 400 mg (KCR 25%) Medium Release
  Arms: NVP ER 400 mg (KCR 25%) Medium Release
Drug: NVP ER 300 mg (KCR 40%) Slow Release
  Arms: NVP ER 300 mg (KCR 40%) Slow Release
Drug: NVP ER 300 mg (ECR 20%) Fast Release
  Arms: NVP ER 300 mg (ECR 20%) Fast Release
Drug: NVP ER 400 mg (KCR 20%) Medium Release
  Arms: NVP ER 400 mg (KCR 20%) Medium Release
Drug: NVP ER 400 mg (KCR 30%) Slow Release
  Arms: NVP ER 400 mg (KCR 30%) Slow Release
Drug: NVP ER 400 mg (KCR 40%) Slow Release
  Arms: NVP ER 400 mg (KCR 40%) Slow Release
Drug: NVP ER 400 mg (ECR 20%) Fast Release
  Arms: NVP ER 400 mg (ECR 20%) Fast Release
Drug: Nevirapine immediate release (IR) 200 mg
  Arms: Nevirapine IR 1 tablet; Nevirapine IR 2 tablets

SUMMARY:
Study to determine the relative bioavailability of different oral Viramune Extended Release (ER) formulations compared to Viramune® Immediate Release (IR) tablet

ELIGIBILITY:
Inclusion Criteria:

* Healthy males according to the following criteria based upon a complete medical history, including the physical examination, vital signs (Blood Pressure (BP), Pulse Rate (PR)), 12-lead electrocardiogram (ECG), clinical laboratory
* Age ≥18 and Age ≤50 years
* Body Mass Index (BMI) ≥18.5 and BMI ≤29.9 kg/m2
* Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice and the local legislation

Exclusion Criteria:

* Any finding of the medical examination (including BP, PR and ECG) deviating from normal and of clinical relevance
* Any evidence of a clinically relevant concomitant disease
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders of clinical relevance
* Surgery of the gastrointestinal tract (except appendectomy and herniotomy)
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History of relevant orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of relevant allergy/hypersensitivity (including allergy to drug or its excipients)
* Intake of drugs with a long half-life (> 24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
* Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial
* Participation in another trial with an investigational drug within two months prior to administration or during the trial
* Smoker (> 10 cigarettes or > 3 cigars or > 3 pipes/day)
* Inability to refrain from smoking on trial days
* Alcohol abuse (more than 60 g/day)
* Drug abuse
* Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
* Excessive physical activities (within one week prior to administration or during the trial)
* Any laboratory value outside the reference range that is of clinical relevance
* Inability to comply with dietary regimen of trial site
* A marked baseline prolongation of QT/QTc interval (e.g., repeated demonstration of a corrected QT interval (QTc) >450 ms)
* A history of additional risk factors for torsade de pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome)
* History of disease which affects the present situation

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 204 (Actual)
Dates: Start 2006-04; Primary Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | up to 144 hours post-dose
Cmax (maximum measured concentration of the analyte in plasma) | up to 144 hours post-dose
C24 (measured concentration of the analyte in plasma at 24 hours post-dose) | 24 hours post-dose

SECONDARY OUTCOMES:
Cmax/C24 ratio | up to 144 hours post-dose
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the time of the last quantifiable data point) | up to 144 hours post-dose
λz (terminal rate constant in plasma) | up to 144 hours post-dose
t1/2 (terminal half-life of the analyte in plasma) | up to 144 hours post-dose
MRTpo (mean residence time of the analyte in the body after po administration) CL/F (apparent clearance of the analyte in the plasma after extravascular administration) | up to 144 hours post-dose
Vz/F (apparent volume of distribution during the terminal phase λz following an extravascular dose) | up to 144 hours post-dose
ka (absorption rate constant) | up to 144 hours post-dose
Number of patients with adverse events | up to 36 days
Assessment of tolerability by investigator on a 4-point scale | within 8 days after last trial procedure
tmax (time from dosing to the maximum concentration of the analyte in plasma) | up to 144 hours post-dose